CLINICAL TRIAL: NCT01997125
Title: Reanimation in Tetraplegia: Restoring Cortical Control of Functional Movement in Humans With Quadriplegia
Brief Title: Reanimation in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marcia Bockbrader (Other)
Responsible Party: Sponsor-Investigator, Marcia Bockbrader, MD, PhD, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013H0164; 2013H0164 (Other: Ohio State University Biomedical IRB)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injury (Quadraplegia)
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Neural bridge system implant and external stimulator
  Interventions: Device: Neural Bridge System

INTERVENTIONS:
Device: Neural Bridge System — Implanted device
  Other Names: Blackrock Microsystems Neuroport; Neuromuscular Stimulator

SUMMARY:
The purpose of this clinical study is to allow the investigation of the Neural Bridging System for participants with tetraplegia to assess if the investigational device can reanimate a paralyzed limb under voluntary control by the participant's thoughts.

DETAILED DESCRIPTION:
This study plans to enroll participants who have been diagnosed with C4- C6 ASIA A spinal cord injuries (motor and sensory complete neurologic injuries), who are more than 1 year post injury, and who are neurologically stable.

ELIGIBILITY:
Inclusion Criteria:

* Must be 21 years or older.
* Must be tetraplegic (C4- C6 ASIA A).
* 12 months post injury and neurologically stable.
* Participant is willing to comply with all follow-up evaluations at the specified times.
* Participant is able to provide informed consent prior to enrollment in the study.
* The participant is fluent in English.
* Participant must have a caregiver willing to participate in the study who will provide care for the surgical site.

Exclusion Criteria:

* No active wound healing or skin breakdown issues.
* No history of poorly controlled autonomic dysreflexia.
* Medical contraindications for general anesthesia, craniotomy, or surgery.
* Diagnosis of acute myocardial infarction or cardiac arrest within previous 6 months.
* Participants with any type of destruction and/or damage to the motor cortex region as determined by MRI.
* History of psychiatric disturbance or dementia
* Other implantable devices such as heart/brain pacemakers
* Participants who rely on ventilators
* Co-morbid conditions that would interfere with study activities or response to treatment.
* History of a neurological ablation procedure.
* Labeled contraindication for MRI.
* History of hemorrhagic stroke.
* History of HIV infection or ongoing chronic infection (such as tuberculosis).
* Pregnant or of child-bearing potential and are not taking acceptable methods of contraception.
* Participation in another FDA device or medication trial that would interfere with the current study.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Bockbrader, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center - Center for Neuromodulation, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bouton CE, Shaikhouni A, Annetta NV, Bockbrader MA, Friedenberg DA, Nielson DM, Sharma G, Sederberg PB, Glenn BC, Mysiw WJ, Morgan AG, Deogaonkar M, Rezai AR. Restoring cortical control of functional movement in a human with quadriplegia. Nature. 2016 May 12;533(7602):247-50. doi: 10.1038/nature17435. Epub 2016 Apr 13. PMID 27074513
- [Result] Sharma G, Friedenberg DA, Annetta N, Glenn B, Bockbrader M, Majstorovic C, Domas S, Mysiw WJ, Rezai A, Bouton C. Using an Artificial Neural Bypass to Restore Cortical Control of Rhythmic Movements in a Human with Quadriplegia. Sci Rep. 2016 Sep 23;6:33807. doi: 10.1038/srep33807. PMID 27658585
- [Result] Friedenberg DA, Bouton CE, Annetta NV, Skomrock N, Mingming Zhang, Schwemmer M, Bockbrader MA, Mysiw WJ, Rezai AR, Bresler HS, Sharma G. Big data challenges in decoding cortical activity in a human with quadriplegia to inform a brain computer interface. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3084-3087. doi: 10.1109/EMBC.2016.7591381. PMID 28268963
- [Result] Friedenberg DA, Schwemmer MA, Landgraf AJ, Annetta NV, Bockbrader MA, Bouton CE, Zhang M, Rezai AR, Mysiw WJ, Bresler HS, Sharma G. Neuroprosthetic-enabled control of graded arm muscle contraction in a paralyzed human. Sci Rep. 2017 Aug 21;7(1):8386. doi: 10.1038/s41598-017-08120-9. PMID 28827605
- [Result] Colachis SC 4th, Bockbrader MA, Zhang M, Friedenberg DA, Annetta NV, Schwemmer MA, Skomrock ND, Mysiw WJ, Rezai AR, Bresler HS, Sharma G. Dexterous Control of Seven Functional Hand Movements Using Cortically-Controlled Transcutaneous Muscle Stimulation in a Person With Tetraplegia. Front Neurosci. 2018 Apr 4;12:208. doi: 10.3389/fnins.2018.00208. eCollection 2018. PMID 29670506
- [Result] Annetta NV, Friend J, Schimmoeller A, Buck VS, Friedenberg DA, Bouton CE, Bockbrader MA, Ganzer PD, Colachis Iv SC, Zhang M, Mysiw WJ, Rezai AR, Sharma G. A High Definition Noninvasive Neuromuscular Electrical Stimulation System for Cortical Control of Combinatorial Rotary Hand Movements in a Human With Tetraplegia. IEEE Trans Biomed Eng. 2019 Apr;66(4):910-919. doi: 10.1109/TBME.2018.2864104. Epub 2018 Aug 7. PMID 30106673
- [Result] Schwemmer MA, Skomrock ND, Sederberg PB, Ting JE, Sharma G, Bockbrader MA, Friedenberg DA. Meeting brain-computer interface user performance expectations using a deep neural network decoding framework. Nat Med. 2018 Nov;24(11):1669-1676. doi: 10.1038/s41591-018-0171-y. Epub 2018 Sep 24. PMID 30250141
- [Result] Skomrock ND, Schwemmer MA, Ting JE, Trivedi HR, Sharma G, Bockbrader MA, Friedenberg DA. A Characterization of Brain-Computer Interface Performance Trade-Offs Using Support Vector Machines and Deep Neural Networks to Decode Movement Intent. Front Neurosci. 2018 Oct 24;12:763. doi: 10.3389/fnins.2018.00763. eCollection 2018. PMID 30459542
- [Result] Bockbrader M, Annetta N, Friedenberg D, Schwemmer M, Skomrock N, Colachis S 4th, Zhang M, Bouton C, Rezai A, Sharma G, Mysiw WJ. Clinically Significant Gains in Skillful Grasp Coordination by an Individual With Tetraplegia Using an Implanted Brain-Computer Interface With Forearm Transcutaneous Muscle Stimulation. Arch Phys Med Rehabil. 2019 Jul;100(7):1201-1217. doi: 10.1016/j.apmr.2018.07.445. Epub 2019 Mar 20. PMID 30902630
- [Derived] Colachis SC 4th, Dunlap CF, Annetta NV, Tamrakar SM, Bockbrader MA, Friedenberg DA. Long-term intracortical microelectrode array performance in a human: a 5 year retrospective analysis. J Neural Eng. 2021 Aug 23;18(4). doi: 10.1088/1741-2552/ac1add. PMID 34352736
- [Derived] Ganzer PD, Colachis SC 4th, Schwemmer MA, Friedenberg DA, Dunlap CF, Swiftney CE, Jacobowitz AF, Weber DJ, Bockbrader MA, Sharma G. Restoring the Sense of Touch Using a Sensorimotor Demultiplexing Neural Interface. Cell. 2020 May 14;181(4):763-773.e12. doi: 10.1016/j.cell.2020.03.054. Epub 2020 Apr 23. PMID 32330415
- [Derived] Zhang M, Schwemmer MA, Ting JE, Majstorovic CE, Friedenberg DA, Bockbrader MA, Jerry Mysiw W, Rezai AR, Annetta NV, Bouton CE, Bresler HS, Sharma G. Extracting wavelet based neural features from human intracortical recordings for neuroprosthetics applications. Bioelectron Med. 2018 Jul 31;4:11. doi: 10.1186/s42234-018-0011-x. eCollection 2018. PMID 32232087

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited 2013-2015 from a tertiary care center rehabilitation clinic
Groups:
- Neural Bridge System - Open Label: Neural bridge system implant and external stimulator
  Neural Bridge System: Implanted device
Period: Overall Study
Arm/Group | Neural Bridge System - Open Label
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neural Bridge System - Open Label
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Number of participants with voluntary movement [Count of Participants; unit: Participants] — Qualitative observation of ability to consistently control hand movement, at baseline without the neural bridge system
  Participants
    Evoked movement - able | 0
    Evoked movement - unable | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Voluntary Movement
Description: The primary outcome measure of this study is the achievement of voluntary hand movement using the neural bridge system
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neural Bridge System - Open Label
Number analyzed (Participants) | 1
Participants
  Voluntary Movement - able | 1
  Voluntary Movement - unable | 0

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term, please consider making this explicit in the Adverse Event Reporting Description
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=1)
Unanticipated, device-related SAE (General disorders) | 1 (1) — Change in psychological sense of self to include functions enabled by use of the neural bridge system, resulting in the participant keeping the neuroimplant (declining explant) at the completion of the study term - deemed a UPIRSO by the study IRB.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=1)
Non-device related AE associated with spinal cord injury (anticipated) (Skin and subcutaneous tissue disorders) | 1 (1) — Complications of deep tissue injury
Non-device related AE associated with spinal cord injury (anticipated) (Renal and urinary disorders) | 1 (1) — Urinary tract infection and bladder stones associated with neurogenic bladder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT01997125/Prot_SAP_000.pdf